CLINICAL TRIAL: NCT07368725
Title: Correlation Study of the Effect of Humeral Tuberosity Fractures on Rotator Cuff Function
Brief Title: The Research About the Function of the Rotator Cuff After Humeral Greater Tuberosity Fractures
Status: Completed | Type: Observational
Sponsor: Guo Jialiang (Other)
Responsible Party: Sponsor-Investigator, Guo Jialiang, Clinical Professor, Hebei Medical University Third Hospital
Organization: Hebei Medical University Third Hospital (Other)
Other Study IDs: GJL002
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff
Keywords: Rotator Cuff Injuries; Rotator Cuff Tears; Humerus Fractures; supraspinatus muscle; infraspinatus muscle
MeSH Terms: conditions — Rotator Cuff Injuries; Humeral Fractures | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated conservatively: All patients had a combined humeral tuberosity fracture with rotator cuff injury, all had CT data, and were treated conservatively
  Interventions: Other: without intervention
- Patients treated surgically: All patients had a combined greater tuberosity humerus fracture with rotator cuff injury, all had CT data, and were treated surgically
  Interventions: Other: without intervention

INTERVENTIONS:
Other: without intervention — without intervention,just retrospectively review the data about patients

SUMMARY:
The purpose of this retrospective study was to investigate the differences in fracture block and rotator cuff function in patients with rotator cuff injuries due to greater tuberosity humerus fractures. Some patients with combined humeral tuberosity fracture and rotator cuff injury can achieve better fracture healing with preservation of acceptable rotator cuff function after 6 months of conservative treatment and rehabilitation. However, other patients require surgery to improve rotator cuff function and relieve shoulder pain and other complications. In this study, two types of patients were followed up at different time points to find out the change of rotator cuff function of the patients. In addition, this study will measure the data related to the fracture bone block on a three-dimensional model created using CT, by which obtaining more accurate measurements than two-dimensional.

ELIGIBILITY:
Inclusion Criteria:

* Three dimensional construction with mimics(with CT of B30);
* Patients older then 18 years;
* Fracture of the greater tuberosity of the humerus combined with rotator cuff injury

Exclusion Criteria:

* Patients with the presence of neurological disease;
* Open fracture;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fracture of the greater tuberosity of the humerus combined with rotator cuff injury
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
classification based on Neer | 2019.01-2024.8

CONTACTS AND LOCATIONS:
Overall Officials: jialiang Guo, Doctor, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- the Third Hospital of Hebei Medical University, Shijiazhuang, Heibei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: after the experiment was conducted
Access Criteria: all authors focusing on rotator cuff